CLINICAL TRIAL: NCT00851201
Title: Comprehensive Approach to Family Weight Management
Brief Title: Family Weight Management Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R18DK075981 (NIH)
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Diabetes
Keywords: children; obesity; weight loss; prevention; diabetes risk; cardiometabolic
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Intervention (Active Comparator)
  Interventions: Behavioral: Standard intervention
- Intensive lifestyle (Experimental)
  Interventions: Behavioral: Intensive lifestyle

INTERVENTIONS:
Behavioral: Intensive lifestyle — The intensive lifestyle intervention will include the standard intervention plus 1)12 core group modules for parents (to address roles and skills) and for children (to enhance motivation and skills and to provide physical activity), 3) Tailored support using a "toolbox" approach from community health workers as extensions of the Family Weight Management professional education staff, and 4) monthly after-core follow-up groups.
  Arms: Intensive lifestyle
Behavioral: Standard intervention — The Standard Intervention will receive: 1) an initial consult, which includes an overview of lifestyle goals, 2) quarterly follow-up, 3) and a monthly newsletter.
  Arms: Standard Intervention

SUMMARY:
The purpose of this study is to address the Healthy People 2010 obesity prevention objective. This study will test the effects of a comprehensive family weight management program on the BMI z-score of 7-12 year-old children with a BMI > 85th percentile who receive primary care in a large municipal Bronx hospital. The intervention framework will draw on social marketing theory and the transtheoretical model of behavioral change to incorporate successful obesity prevention strategies. A two-arm randomized controlled clinical trial (RCT), which will enroll (n =506) 7-12 year old children with a > 85th BMI percentile, will compare the Experimental Intensive Intervention to a Standard (Control) Intervention. The Standard Intervention will receive: 1) an initial consult, which includes an overview of lifestyle goals, 2)quarterly follow-up, 3) and a monthly newsletter. The Intensive Intervention will add: 1)12 core group modules for parents (to address roles and skills) and for children (to enhance motivation and skills and to provide physical activity), 3) Tailored support using a "toolbox" approach from community health workers as extensions of the Family Weight Management professional education staff, and 4) monthly after-core follow-up groups. The study will determine if children randomized to the Experimental Intensive Intervention will have greater improvement in BMI change (z-scores) than those randomized to the Control Standard Intervention. The study will also evaluate the effects on the Experimental Intervention on lifestyle variables and assess intervention costs. The RE-AIM evaluation will address: Reach: How many of the eligible children/ families were referred and how many of those referred actually enrolled? We will use BMI data in the computerized medical records to evaluate the proportion and the appropriateness of the referrals. Efficacy/Effectiveness: How did the Experimental intervention affect BMI (changes in z-score), and key biomarkers when followed as planned? Adoption: How acceptable were the intervention(s) to the primary care medical team and the children/families in the pediatric clinics etc? (from process measures and post intervention surveys) Implementation: How many of the intervention activities were provided as planned? Quality control measures will be used to evaluate the integrity of the intervention(s). Maintenance: How much of the intervention effect is sustainable? Individual effects will be evaluated based on the 24 month follow data. Institutional effects evaluation will include the potential to maintain services using third-party coverage.

ELIGIBILITY:
Inclusion Criteria:

BMI greater than 85th percentile for sex, age 7-12 years

Exclusion Criteria:

health or condition that would interfere with study participation, unwilling or inability to provide parent/guardian consent or child ascent, intention to move from area

-

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2009-08; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
BMI percentile for age and sex, biomarkers e.g, glucose, insulin, lipids | 12 months after randomization

SECONDARY OUTCOMES:
dietary intake, and physical activity measures | 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Judith Wylie-Rosett, EdD, RD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- North Bronx Health Network, The Bronx, New York, United States

REFERENCES:
- [Background] Wylie-Rosett J, Isasi C, Soroudi N, Soroker E, Sizemore C, Groisman-Perelstein A, Bass J, Diamantis P, Ahmed T, Gandhi R. KidWAVE: Get Healthy Game--promoting a more healthful lifestyle in overweight children. J Nutr Educ Behav. 2010 May-Jun;42(3):210-2. doi: 10.1016/j.jneb.2009.12.003. No abstract available. PMID 20434077
- [Background] Wright ND, Groisman-Perelstein AE, Wylie-Rosett J, Vernon N, Diamantis PM, Isasi CR. A lifestyle assessment and intervention tool for pediatric weight management: the HABITS questionnaire. J Hum Nutr Diet. 2011 Feb;24(1):96-100. doi: 10.1111/j.1365-277X.2010.01126.x. Epub 2010 Sep 30. PMID 21210873
- [Derived] Matthan NR, Wylie-Rosett J, Xue X, Gao Q, Groisman-Perelstein AE, Diamantis PM, Ginsberg M, Mossavar-Rahmani Y, Barger K, Lichtenstein AH. Effect of a Family-Based Intervention on Nutrient Biomarkers, Desaturase Enzyme Activities, and Cardiometabolic Risk Factors in Children with Overweight and Obesity. Curr Dev Nutr. 2019 Dec 2;4(1):nzz138. doi: 10.1093/cdn/nzz138. eCollection 2020 Jan. PMID 31922084
- [Derived] Wylie-Rosett J, Groisman-Perelstein AE, Diamantis PM, Jimenez CC, Shankar V, Conlon BA, Mossavar-Rahmani Y, Isasi CR, Martin SN, Ginsberg M, Matthan NR, Lichtenstein AH. Embedding weight management into safety-net pediatric primary care: randomized controlled trial. Int J Behav Nutr Phys Act. 2018 Jan 22;15(1):12. doi: 10.1186/s12966-017-0639-z. PMID 29357894
- [Derived] Khan UI, McGinn AP, Isasi CR, Groisman-Perelstein A, Diamantis PM, Ginsberg M, Wylie-Rosett J. Differences in Cardiometabolic Risk between Insulin-Sensitive and Insulin-Resistant Overweight and Obese Children. Child Obes. 2015 Jun;11(3):289-96. doi: 10.1089/chi.2014.0112. Epub 2015 Mar 16. PMID 25774664